CLINICAL TRIAL: NCT06420934
Title: Comparison of the Breach of the Aseptic Barrier After Surgical Handwashing: Drying With One or Two Surgical Towels
Brief Title: Surgical Handwashing: Drying With One or Two Surgical Towels
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Ortopedia Infantil Roosevelt (Other)
Collaborators: Hospital Universitario San Ignacio (Other); Hospital Militar Central, Argentina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2022121502-001
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Hand Hygiene; Surgical Wound Infection; Healthcare Associated Infection; Medical Errors
Keywords: Surgical Scrubbing; Handwashing; Disinfection; Healthcare Associated Infection; Hand Hygiene
MeSH Terms: conditions — Surgical Wound Infection; Cross Infection

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Masking will be provided to data analysis expert.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One surgical towel (Active Comparator): Participants will be asked to remove all accessories from the forearm, wrist, fingers and to roll up any clothing until at least 5 cm above the humeral condyles are exposed. They will be instructed to perform conventional surgical scrubbing and to dry their hands with a conventional paper towel. The research assistant will open the opaque envelope, which will indicate that the participant needs to dry their hands with one surgical towel.
  Interventions: Other: Drying procedure after surgical handwashing
- Two surgical towel (Experimental): Participants will be asked to remove all accessories from the forearm, wrist, fingers and to roll up any clothing until at least 5 cm above the humeral condyles are exposed. They will be instructed to perform conventional surgical scrubbing and to dry their hands with a conventional paper towel. The research assistant will open the opaque envelope, which will indicate that the participant needs to dry their hands with two surgical towels, one for each hand.
  Interventions: Other: Drying procedure after surgical handwashing

INTERVENTIONS:
Other: Drying procedure after surgical handwashing — Participants will dry their hands with one surgical towel

SUMMARY:
This study aims to determine whether the use of two sterile towels for drying after surgical handwashing results in fewer contamination events compared to the use of only one towel among healthcare personnel. This randomized, multicenter, superiority-controlled trial will enroll up to 72 healthcare workers and surgical residents from three hospitals in Bogotá, Colombia. A fluorescent product will simulate bacteria, and contamination will be assessed by evaluating the presence of fluorescent cream after hand drying technique with either two or one surgical sterile towel. Data will be collected through REDCap and deidentified. Differences in the proportion of contamination between the two groups will be assessed using an exact Fischer test, and confounding variables will be included in the analysis through logistic multivariate regression, with a significance level set a priori at 0.05. Results will be submitted for publication in a peer-reviewed journal.

DETAILED DESCRIPTION:
Approval was obtained from the ethics committee of three healthcare institutions. A process of informed consent will be conducted with all participants, and confidentiality and data protection will be guaranteed. A research assistant, unaware of the operational hypotheses and study objectives, will execute the experiment and record the results. There will be no blinding of the intervention for the participants or the assistant. At each institution, randomization will be conducted a priori to determine the operating room where participants should be recruited. Likewise, the intervention to be administered will be randomized. All these data will be stored in opaque envelopes that will be opened at the time of recruitment. A total of 72 participants will be recruited, with 36 exposed to drying with one towel and 36 to drying with two towels. Recruitment will cease upon completion of the respective participants stipulated for each intervention.

The primary outcome of interest will be the presence or absence of contamination. To evaluate this outcome, the gold standard would be the collection of cultures and the analysis of the presence or absence of bacterial contamination. However, due to the costs and methodological difficulties of taking cultures, an indirect method, previously validated as a surrogate, will be employed instead. 2 mL of fluorescent cream (Glo Germ ™) will be applied with a brush proximal to the normally washed area during surgical scrubbing (3 cm above the elbow). Participants will be shown a video on how to dry with one or two surgical towels and will be given one minute to do so. Subsequently, the presence or absence of fluorescent cream on the upper extremities will be evaluated using a UV light lamp. If fluorescence is evidenced in the washed area where it was not applied, it will be considered that there was contamination during the hand drying process.

No interim analyses will be executed. Data will be de-identified for the analysis. Descriptive statistics will be conducted using R studio, and proportions of contamination when drying with one or two towels will be compared. A simple logistic regression will be performed to assess the relationship between the intervention and the proportion of contamination events, and a multivariate logistic regression will be conducted to assess the effect of confounding variables on the outcome. The results will be reported collectively for publication in a peer-reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* Workers and students who have a current affiliation with the institutions where the study will be executed.
* Workers and students whose practice or work involves performing surgical handwashing at least once a week for invasive procedures.

Exclusion Criteria:

* Workers and students who do not wish to participate in the study.
* Workers and students whose work activities do not allow them time to participate in the study.
* Workers and students who are allergic to the fluorescent cream
* Workers and students whose nails exceed a length of 0.5 cm from the fingertip edge.
* Workers and students whose nails are painted with polish.
* Workers and students who refuse to remove jewelry and accessories from wrists and hands.
* Workers and students with recent wounds on hands or forearms, including tattoos done in the last month.
* Workers and students who do not adhere to the handwashing and drying technique taught prior to the study's implementation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Contamination | 3 minutes after handwash and hand drying.
  Presence or absence of fluorescent cream on the upper extremities will be evaluated using a UV light lamp in a dark room. If fluorescence is observed in the washed area where it was not applied, it will be considered that there was contamination during the hand drying process.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Ortopedia Infantil Roosevelt, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WHO Guidelines on Hand Hygiene in Health Care: First Global Patient Safety Challenge Clean Care Is Safer Care. Geneva: World Health Organization; 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK144013/ PMID 23805438
- [Background] Nicolay CR. Hand hygiene: an evidence-based review for surgeons. Int J Surg. 2006;4(1):53-65. doi: 10.1016/j.ijsu.2005.06.002. Epub 2005 Aug 1. PMID 17462314
- [Background] Huang C, Ma W, Stack S. The hygienic efficacy of different hand-drying methods: a review of the evidence. Mayo Clin Proc. 2012 Aug;87(8):791-8. doi: 10.1016/j.mayocp.2012.02.019. Epub 2012 May 31. PMID 22656243
- [Background] Gustafson DR, Vetter EA, Larson DR, Ilstrup DM, Maker MD, Thompson RL, Cockerill FR 3rd. Effects of 4 hand-drying methods for removing bacteria from washed hands: a randomized trial. Mayo Clin Proc. 2000 Jul;75(7):705-8. doi: 10.4065/75.7.705. PMID 10907386
- [Background] Suen LKP, Lung VYT, Boost MV, Au-Yeung CH, Siu GKH. Microbiological evaluation of different hand drying methods for removing bacteria from washed hands. Sci Rep. 2019 Sep 24;9(1):13754. doi: 10.1038/s41598-019-50239-4. PMID 31551459
- [Background] Mutters R, Warnes SL. The method used to dry washed hands affects the number and type of transient and residential bacteria remaining on the skin. J Hosp Infect. 2019 Apr;101(4):408-413. doi: 10.1016/j.jhin.2018.12.005. Epub 2018 Dec 8. PMID 30537524
- [Background] Handaya AY, Werdana VAP. Adherence to preoperative hand hygiene and sterile gowning technique among consultant surgeons, surgical residents, and nurses: a pilot study at an academic medical center in Indonesia. Patient Saf Surg. 2019 Mar 11;13:11. doi: 10.1186/s13037-019-0193-5. eCollection 2019. PMID 30899331
- [Background] Skodova M, Garcia Urra F, Gimeno Benitez A, Jimenez Romano MR, Gimeno Ortiz A. Hand hygiene assessment in the workplace using a UV lamp. Am J Infect Control. 2015 Dec 1;43(12):1360-2. doi: 10.1016/j.ajic.2015.07.003. Epub 2015 Aug 18. PMID 26297523
- [Background] Szilagyi L, Lehotsky A, Nagy M, Haidegger T, Benyo B, Benyo Z. Stery-hand: A new device to support hand disinfection. Annu Int Conf IEEE Eng Med Biol Soc. 2010;2010:4756-9. doi: 10.1109/IEMBS.2010.5626377. PMID 21096021
- [Background] Sakmen KD, Sterz J, Stefanescu MC, Zabel J, Lehmann M, Ruesseler M. Impact of the teaching method of the rub-in technique for learning hygienic hand disinfection in medical studies: a comparative effectiveness analysis of two techniques. GMS Hyg Infect Control. 2019 Nov 13;14:Doc17. doi: 10.3205/dgkh000332. eCollection 2019. PMID 31815090
- [Background] Marena C, Lodola L, Zecca M, Bulgheroni A, Carretto E, Maserati R, Zambianchi L. Assessment of handwashing practices with chemical and microbiologic methods: preliminary results from a prospective crossover study. Am J Infect Control. 2002 Oct;30(6):334-40. doi: 10.1067/mic.2002.125809. PMID 12360141